CLINICAL TRIAL: NCT05880238
Title: The Effect of Occupational Therapy-Based Sensory Motor Training On Self-Regulation, Cognitive Skills, And School Readiness in Preschool Children
Brief Title: The Effect of Sensory Motor Training in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Remziye Akarsu, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pre-school intervention
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Early Intervention
Keywords: pre-school; sensory-motor; self-regulation; school readiness
MeSH Terms: conditions — Self-Control | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory-motor training (Experimental): The study group received group interventions that included self-regulation strategies and sensory-motor skill training in addition to preschool education. Group interventions were conducted with groups of up to 10 participants for a total of one hour, twice a week for 10 weeks.
  Interventions: Behavioral: Intervention group
- Control (Active Comparator): The control group continued with preschool education and did not receive any additional intervention.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Intervention group — The intervention consisted of a total of 3 modules, 20 sessions. These modules are: Module A: I explore my inner and outer world Module B: I am learning self-editing methods C module: discovering self-editing In these modules, students were trained to use sensorimotor strategies for self-regulation. The intervention program was carried out in one-hour sessions, twice a week, for a total of 10 weeks.
  Arms: Sensory-motor training
Other: Control group — The control group will continue their education according to the preschool education curriculum.
  Arms: Control

SUMMARY:
When looking at the literature, sensory-motor skills, self-regulation, executive functions, cognitive styles, and school readiness are strongly related concepts. Self-regulation skills are closely related to the maturity of sensory-motor components. Therefore, it is important to provide sensory-motor training with self-regulation strategies. However, no study investigating the effects of self-regulation strategies combined with sensory-motor training on school readiness, self-regulation, executive functions, and cognitive styles could be found in the literature.

Our study aims to examine the effect of self-regulation strategies and occupational therapy-based sensory-motor training on self-regulation, cognitive skills, and school readiness in preschool children.

The research will be carried out in two preschool classrooms of students aged 5-6 years registered for the 2022-2023 academic year at Özel Mavi Umut Eğitim Kurumları in Istanbul.

A total of 38 children will participate in the study, 19 in the intervention group and 19 in the control group. While the control group continues their preschool education, the intervention group will receive group interventions including self-regulation strategies and sensory-motor skills training for 1 hour, twice a week, for 10 weeks, in addition to their regular preschool education.

Metropolitan School Readiness Test, Kansas Pre-School Self-Concept Scale Form A, Childhood Executive Function Inventory, Pre-School Self-Regulation Scale, Dunn Sensory Profile, and Bruininks-Oseretsky Short Form 2 will use to evaluate both the intervention and control groups at 10-week intervals.

The data obtained from the evaluations will be analyzed using SPSS (Statistical Package for Social Science) 22.0 version. If the data follows a normal distribution, the Paired Student's t-test will be used for comparison, and if not, the Wilcoxon Matched Two-Sample Test will be used. Mean±standard deviation (X±SD) will be determined for the identified variables. A statistical significance level of p≤0.05 will be considered.

DETAILED DESCRIPTION:
The purpose of our study is to investigate the effect of self-regulation strategies and occupational therapy-based sensory-motor education on self-regulation, cognitive skills, and school readiness in preschool children.

The research will be carried out in two kindergarten classes consisting of students aged 5-6 years, registered as part of the 2022-2023 academic year at Özel Mavi Umut Eğitim Kurumları located in Istanbul. In the G-Power program, based on the literature information, it was calculated that at least 15 people should participate in the study for each group, considering the values of 1.33±1.27 (mean±SD difference between groups) for 95% power (Fathirezaie et al., 2021). A total of 38 children, including 19 children whom will receive self-regulation strategies and a sensory-motor education program in the study group and 19 children in the control group, will include in the study.

To sustain the experimental study, an easily accessible preschool institution was selected. Kindergarten classes at Özel Mavi Umut Eğitim Kurumları will determine as the study and control group using a simple random sampling method.

While the control group continues preschool education, group interventions, including self-regulation strategies and sensory-motor skill training, will be applied to the study group in addition to preschool education. Group interventions will be conducted twice a week for a total of one hour for 10 weeks, with groups consisting of up to 10 people.

The inclusion criteria were attending preschool education, being between the ages of 5-6, and not having started primary school. Children with neurological, orthopedic, psychiatric diagnoses, and sensory impairments (e.g. visual and hearing loss) were excluded from the study.

EVALUATION TOOLS Parent-child information form (including questions that comply with inclusion criteria and general demographic information such as body mass index and education)

Primary outcome measures

Metropolitan School Readiness Test: Developed by G.H. Hildreth, N.L. Griffiths, and M. Mc Gauvran in 1949, this test was adapted into Turkish by Oktay (1980) and is used to measure the characteristics that determine the school readiness and the level of school readiness of children who are starting school. The test consists of two sub-dimensions: reading readiness and number readiness, and a total of 100 items. The reading readiness sub-dimension consists of 66 items, including word comprehension (19), sentences (14), general knowledge (14), and matching (19). The number readiness sub-dimension consists of 34 items, including numbers (24) and copying (10) (Oktay, 1983, p. 35). In the reliability study carried out within this scope, the correlations between parallel forms applied at certain intervals to 195 first-grade students were calculated, and the reliability coefficients obtained were found to range from .53 to .83. American norms and Istanbul norms were compared for the validity of the test. In the study, the test was applied to children living in certain regions of Istanbul and compared with the American norms.

The Kansas Reflection-Impulsivity Scale for Preschool Children A Form (KRISP) is a scale developed by Wright (1971) to determine children's cognitive tempo. The scale consists of 10 shapes and 5 example shapes that will be used to teach children how to apply the scale. The validity and reliability studies of the scale were conducted by Seçer et al. (2010). For the scope and face validity of the scale, expert opinions were obtained. For reliability studies, scorer reliability, test-retest, and split-half reliability were preferred. For scorer reliability, 30 six-year-old students were evaluated by two different observers for response time. The correlation between the two observers was found to be r = 0.83 for response time and r = 0.78 for error rate. Test-retest reliability was examined by selecting a study group of 303 children attending preschool education institutions in the center of Konya and applying the scale twice with a two-week interval, and Pearson's Moment Correlation Coefficient was examined between application scores. The correlation coefficient was r = 0.74 for error rate and r = 0.89 for response time. There was a positive, significant (p <.01) relationship between the two separate applications in the same group. As a result of the findings, it was concluded that the consistency between the two applications of the scale was at an acceptable level. To determine the reliability of the test, the split-half method was also used. The correlation coefficient calculated using the Spearman-Brown formula for response time was r = 0.85, and for error rate was r = 0.71 (Seçer et al., 2010).

The scale is applied one-on-one with the child by the researcher. Before the application, the researcher prepares a note paper where the child's information will be recorded, and the child is taught how to apply the scale using the five example shapes available in the scale. Once the child has learned how to apply the scale, the actual shapes are shown to the child one by one. Pages containing the actual shape and six pages with shapes that are almost identical to the actual shape are shown to the child at the same time, and the child is asked to find the same shape as the actual one among the other six shapes. The timer is started as soon as the instruction is given to the child, and the child's first response time is recorded on the prepared paper. If the answer is correct, the same process is repeated for the other shapes, and if the answer is incorrect, another instruction is given to the child to find the correct shape, and all answers are recorded. The number of mistakes the child makes until finding the correct answer is also noted in this paper.

The Childhood Executive Functioning Inventory (CHEXI) is a measurement tool developed by Thorell and Nyberg (2008) that focuses on the executive functions of children aged 4-12. The questions in the inventory were created based on Barkley's (1997) model, which explains that inhibitory control, working memory, and self-regulation create significant executive function disorders in children with ADHD. Initially, 26 items were categorized into four sub-dimensions. According to this, 11 items were considered "working memory," four items were considered "planning," six items were considered "inhibitory control," and five items were considered "regulation." However, items 25 and 26 were not included in the factor analysis due to very low sample suitability. According to the results of the factor analysis, a two-factor structure provided the best fit to the data: (1) working memory and (2) inhibitory control. The first factor includes the items of working memory and planning sub-dimensions, while the second factor includes the items of inhibitory control and regulation sub-dimensions. In addition, the correlation between the two factors was found to be 0.65. All of these analyses were first performed for the parental form of the inventory. In the study conducted with the teacher form, a two-factor structure also emerged. In teacher evaluations, the correlation between the two factors was found to be 0.69 (Thorell and Nyberg, 2008). As a result, the CDYIE consists of 24 items. Working Memory contains 13 items (e.g., "Has difficulty remembering what they were doing in the middle of an activity"), while Inhibitory Control contains 11 items (e.g., "Has difficulty restraining or controlling oneself even when told to do so"). The scale can be completed by parents or teachers. The scale is a 5-point Likert scale. After each statement, the parent or teacher indicates how true the statement is for the child by circling one of the numbers (1 to 5) provided (1: Not true, 5: True). Filling out the scale takes 5-10 minutes (Thorell and Catale, 2014; Thorell and Nyberg, 2008). High scores on the scale indicate that the child has more difficulties related to executive functions. Therefore, it can be interpreted that children who score lower on the inventory have higher levels of executive functions than those who score higher (Thorell and Nyberg, 2008). However, in this study, all items were reverse-coded to represent an increase in executive function skills rather than difficulties, so higher scores indicate that the child shows more executive function skills.

Secondary Outcome Measures

Dunn Sensory Profile: Sensory Profile, developed by Occupational Therapist Prof. Winnie Dunn, is a measurement tool used to evaluate an individual's tendency to respond to sensory stimuli during daily activities, also known as sensory modulation, and which sensory systems affect daily life more. The validity and reliability of this test have been demonstrated. The test is used to measure an individual's functional performance in daily life activities, sensory processing abilities, and sensory processing impact, and is evaluated based on a Likert scale (1 = Always, 2 = Often, 3 = Sometimes, 4 = Rarely, 5 = Never) with 9-factor scores consisting of 3 main sub-parameters (sensory processing, modulation, and behavioral-emotional responses). Typical performance, possible differences, and definite difference score ranges have been determined for each parameter. As the total score for each parameter progresses towards the typical performance score range from the definite difference score range, improvement is observed (Dunn, 1999). The validity and reliability of the Sensory Profile test have been established (Kayıhan et al., 2012).

Bruininks-Oseretsky Test 2 Short Form: The development of the Bruininks-Oseretsky Motor Proficiency Test (BOMPT) began in 1972 by Robert H. Bruininks based on the Oseretsky Motor Proficiency Test. After six years of work, Dr. Robert H. Bruininks developed the test (Bruininks, 2005; Crowe, 1989). The BOMPT was developed to measure the motor functions of children aged 4.5-14 years. The long form of the BOMPT consists of 8 sub-tests and a total of 46 items. It is also a comprehensive motor proficiency indicator and measures both gross and fine motor skills. In 2005, the Bruininks-Oseretsky Motor Proficiency Test was updated and became the Bruininks-Oseretsky Test 2 (BOT2). BOT2 applies to children aged 4-21 years. The validity and reliability of BOT2 long form were tested on healthy children aged 5 years by Ballı in 2012 (Ballı and Gürsoy, 2012; Bruininks and Oseretsky, 2010). BOT2-KF was updated in 2010. BOT2-KF consists of 8 sub-tests and 12 items in total. The test takes about 15-20 minutes to administer. A person can obtain a maximum of 72 processed points from the test. A Turkish validity and reliability study has been conducted (Köse et al., 2021).

INTERVENTION PROGRAM The study will be conducted as a group intervention for 10 weeks, with each training session lasting one hour, twice a week. The group intervention will be implemented with 10 children in each group.

The control group will continue their preschool education, and the same evaluations will be applied to this group at a 10-week interval.

Existing programs in the literature on self-regulation strategies and sensory-motor education planning will be used in the content of the program.

Assessment tools will be applied to the study and control group children at a 10-week interval. The data obtained from the evaluation will be analyzed using the SPSS (Statistical Package for Social Science) 22.0 version. After checking whether the data conforms to a normal distribution with the Shapiro-Wilk test, if the data is normally distributed, the paired samples Student's t-test will be used for statistical comparison, and if not, the Wilcoxon Matched-Pairs Two-Sample Test will be used. Mean±standard deviation (X±SS) will be determined for the identified variables. A significance level of p≤0.05 will be accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* to attend preschool education class
* to be between the ages of 5-6
* not to have started primary school yet

Exclusion Criteria:

* to have a neurological, orthopedic, or psychiatric diagnosis,
* to have a sensory disability (e.g. visual and hearing loss).

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Metropolitan School Readiness Test | two weeks
  The Metropolitan School Readiness Test was developed by G. H. Hildreth, N. L. Griffits, and M. Mc Gauvran in 1949. This test was adapted into Turkish by Oktay (1980) and is used to measure the characteristics and levels of school readiness for children who are starting school. The test consists of two sub-dimensions: reading readiness and number readiness, and a total of 100 items. The reading readiness sub-dimension consists of 66 items, including word meaning (19), sentences (14), general knowledge (14), and matching (19). The number readiness sub-dimension consists of 34 items, including numbers (24) and copying (10) (Oktay, 1983, p. 35). Higher scores indicate higher performance.
Kansas Reflection-Impulsivity for Preschool-KRISP | one week
  The scale used to determine the cognitive tempo of children is the Form A of the Kansas Reflection-Impulsivity for Preschool-KRISP developed by Wright (1971). The scale consists of 10 shapes and 5 sample shapes that will be used to teach children how to use the scale. Higher scores indicate higher performance.
Childhood Executive Functioning Invantery-CHEXI | one week
  The measurement tool developed by Thorell and Nyberg (2008) focuses on the executive functions of children aged 4-12 years old. The questions in the scale were created based on Barkley's (1997) model, which explains that inhibitory control, working memory, and self-regulation create significant executive function impairments in children with ADHD. The lover scores indicate higher performance.
Preschool Self-Regulation Scale | two weeks
  The Preschool Self-Regulation Assessment (PSRA), developed by Smith-Donald et al. (2007), is a performance-based assessment tool that enables evaluators to assess children's emotions, attention, and behaviors based on practitioner-child interactions. The Practitioner Rating Form in the PSRA is a rubric-style assessment tool that is scored from 0 to 3 based on the items used. The Turkish adaptation of the PSRA was carried out by Ezgi Fındık Tanrıbuyurdu and Güler Yıldız in 2012 (Tanrubuyurdu and Yıldız, 2012). The higher scores indicate higher performance.

SECONDARY OUTCOMES:
Sensory Profile | one week
  The Sensory Profile, developed by Occupational Therapist Prof. Winnie Dunn, is a measurement tool used to evaluate an individual's sensory modulation, or in other words, their tendency to respond to sensory stimuli during daily activities and which sensory systems are most affected. The validity and reliability of this test have been shown. The test is used to measure an individual's functional performance in daily life activities, sensory processing abilities, and sensory processing impact. It consists of three main sub-parameters (sensory processing, modulation, and behavioral-emotional responses) and nine factor scores composed of a Likert scale (1 = Always, 2 = Often, 3 = Sometimes, 4 = Rarely, 5 = Never). Typical performance, potential differences, and definitive difference score ranges have been established for each parameter. As the total score for each parameter approaches the typical performance score range from the definitive difference score range, improvement is seen.
Bruininks-Oseretsky Test 2 Short Form | two weeks
  The BOT2-KF consists of a total of 8 subtests and 12 items. The administration of the test takes approximately 15-20 minutes. A person can receive a maximum of 72 processed points from the test. The validity and reliability study of the test has been conducted in Turkish (Köse et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Remziye Akarsu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No